CLINICAL TRIAL: NCT03049176
Title: The Impact and Cost-effectiveness of Safer Conception Strategies for HIV-discordant Couples
Brief Title: The Impact and Cost-effectiveness of Safer Conception Strategies for HIV-discordant Couples (SAFER)
Acronym: SAFER
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: UZ-UCSF Collaborative Research Programme (Other); National Institute of Mental Health (NIMH) (NIH); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Joelle Brown, MPH, PhD, Principal Investigator, University of California, San Francisco
Other Study IDs: A126763; K01MH100994 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections
Keywords: HIV-discordant couple; ART; PrEP; semen washing; artificial vaginal insemination; safer conception; pregnancy
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Anti-Retroviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV+male/HIV-female: discordant couple given the choice of using at least one of the following: Antiretrovirals, PrEP (Truvada), or semen washing
  Interventions: Drug: PrEP (Truvada); Drug: Antiretrovirals; Procedure: Semen washing
- HIV+female/HIV-male: discordant couple given the choice of using at least one of the following: Antiretrovirals, PrEP (Truvada), or artificial vaginal insemination
  Interventions: Drug: PrEP (Truvada); Drug: Antiretrovirals; Procedure: Artificial vaginal insemination

INTERVENTIONS:
Drug: PrEP (Truvada) — oral, daily Truvada for HIV-negative participants
  Other Names: emtricitabine/tenofovir disoproxil fumarate
Drug: Antiretrovirals — oral daily antiretrovirals and frequent viral load monitoring for HIV-positive participant
  Other Names: ART
Procedure: Semen washing — collection of semen from an HIV-positive man, processing semen to remove HIV, followed by intrauterine insemination
  Groups: HIV+male/HIV-female
Procedure: Artificial vaginal insemination — collection of semen from an HIV-negative man, followed by intravaginal insemination
  Groups: HIV+female/HIV-male

SUMMARY:
This is a prospective, non-randomized, open-label study to look at the uptake, adherence to, and impact of pre-exposure prophylaxis (PrEP), antiretroviral therapy (ART), semen washing, and vaginal insemination to prevent HIV among HIV-discordant couples attempting conception in Zimbabwe.

DETAILED DESCRIPTION:
The reproductive needs of HIV-discordant couples who desire pregnancy represent an urgent public health problem that has been neglected in HIV prevention research. In Zimbabwe , and across sub-Saharan Africa, the vast majority of HIV-infected individuals are adults of reproductive age. Pregnancy and the desire for children are common among HIV-infected individuals, and HIV-discordant couples face a difficult choice between attempting pregnancy and risking HIV transmission to their partners. Recent surveys have found that 30-50% of HIV-infected individuals in sub-Saharan Africa are involved in stable, HIV-discordant relationships, and HIV transmission within married, cohabitating HIV-discordant couples accounts for 44-60% of new HIV infections in some regions of sub-Saharan Africa. While knowledge of HIV discordance can lead to increased condom use, many discordant couples have unprotected intercourse often motivated by the desire to conceive. Currently, HIV discordant couples who attempt to conceive place themselves at considerable risk of transmission. This research study aims to help promote couples' rights to conceive while at the same time decreasing the risk of HIV transmission.

ELIGIBILITY:
Inclusion Criteria:

For all couples:

* Couple expresses a desire to conceive
* Sexually active (defined as having vaginal sex with one another at least 6 times in the past 3 months
* Willing to enter the study as a couple and intending to remain as a couple and have a sexual relationship for the next 12 months
* Willing to use at least one safer conception strategy
* For men, age ≥18 years. For women, age 18 - 35 years;
* Able and willing to provide written informed consent

For HIV-uninfected members of the couple

* HIV-negative based on parallel negative HIV rapid tests, both at study screening and enrollment visit
* Adequate renal function, defined by normal creatinine levels and estimated creatinine clearance ≥60 mL/min

For HIV-infected members of the couple

* HIV-positive based on parallel positive HIV rapid tests, based on national algorithm
* No current AIDS-defining illness

Exclusion Criteria:

* Amenorrheic
* Currently pregnant
* Active and serious infections, including active tuberculosis infection; active clinically significant medical problems including cardiac disease, pulmonary disease, and previously diagnosed malignancy expected to require further treatment.
* History of infertility defined as a year or more of regular unprotected intercourse with current partner without pregnancy, or otherwise medically diagnosed infertility
* Currently on any concomitant medication that requires the participant to avoid use of PrEP

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV-discordant couples in Harare, Zimbabwe who are trying to get pregnant
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Uptake of safer conception strategies | 12 months
  proportion of couples choosing the strategy
Acceptability of safer conception strategies | 12 months
  proportion of couples remaining on strategy; reports of satisfaction
Adherence to safer conception strategies | 12 months
  proportion of couples with high adherence to strategy

SECONDARY OUTCOMES:
Effectiveness of safer conception strategies on HIV prevention | 12 months
  incidence of HIV
Effectiveness of safer conception strategies on achieving pregnancy | 12 months
  incidence of pregnancy
costs of providing safer conception services | 12 months
  costs
cost-effectiveness of safer conception strategies | 12 months
  model the cost effectiveness of various combinations of safer conception strategies

CONTACTS AND LOCATIONS:
Overall Officials: Joelle M Brown, PhD, MPH, Principal Investigator — University of California, San Francisco; Felix Mhlanga, MBChB, MMed, Principal Investigator — UZ-UCSF Collaborative Research Programme
Locations (1):
- UZCHS-UCSF CTRC Zengeza Clinical Research Site, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available at the end of the study on an online repository.

REFERENCES:
- [Derived] Brown JM, Gitome S, Mataveke B, Chirenda T, Matubu A, Chareka G, Chasakara C, Mgodi N, Murombedzi C, Musara P, Makurumure T, Hughes CS, Bukusi E, Cohen CR, Shiboski S, Darbes L, Kahn JG, Rutherford GW, Chirenje ZM, Mhlanga F. Preventing HIV and achieving pregnancy among HIV sero-different couples: Pilot study of a safer conception intervention in Zimbabwe. PLOS Glob Public Health. 2023 Feb 24;3(2):e0000796. doi: 10.1371/journal.pgph.0000796. eCollection 2023. PMID 36963004
- [Derived] Hughes CS, Brown J, Murombedzi C, Chirenda T, Chareka G, Mhlanga F, Mateveke B, Gitome S, Makurumure T, Matubu A, Mgodi N, Chirenje Z, Kahn JG. Estimated costs for the delivery of safer conception strategies for HIV-discordant couples in Zimbabwe: a cost analysis. BMC Health Serv Res. 2020 Oct 12;20(1):940. doi: 10.1186/s12913-020-05784-4. PMID 33046066